CLINICAL TRIAL: NCT04619082
Title: The Efficacy and Safety of TAF as a Prophylactic Antiviral Agent for HBsAg-positive Cancer Patients Receiving Chemotherapy
Brief Title: TAF to Prevent HBV Reactivation in Cancer Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Collaborators: St. Martin De Porress Hospital (Other); Dalin Tzu Chi General Hospital (Other); National Taiwan University Hospital, Yun-Lin Branch (Other); Chi Mei Medical Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB2020091
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B Reactivation
Keywords: TAF; cancer patients; chemotherapy
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAF prophylaxis (Experimental): Using TAF to prevent HBV reactivation for HBsAg-positive cancer patients
  Interventions: Drug: Tenofovir alafenamide

INTERVENTIONS:
Drug: Tenofovir alafenamide — Tenofovir alafenamide 25 mg once per day for one year

SUMMARY:
Tenofovir alafenamide (TAF) has been approved to prevent HBV reactivation for HBsAg-positive cancer patients receiving chemotherapy. However, the real-world effectiveness and safety of TAF for cancer patients was lacing. Therefore, we conduct a prospective single arm study to evaluate the efficacy and safety of TAF as a prophylactic antiviral agent for HBsAg-positive cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
This prospective single arm study would be conducted in Taiwan. Patients who fulfill the inclusion criteria, will receive TAF before the initiation of systemic chemotherapy. Based on the guidance of NHI in Taiwan, prophylactic anti-viral agent should be prescribed within 7 days before chemotherapy and would be discontinued at 6 months after cessation of chemotherapy. The duration of TAF prophylaxis would be followed the guidance of NHI in Taiwan, however, the end of our observation would be at week 48 after TAF use. Patients will receive regular follow up at week 4, 12, 24, 36 and 48 (for T-bil, AST, ALT, creatinine, HBsAg, HBV DNA) till 1 year and the outcome will be collected. Platelet and HBcrAg would be examined at enrollment, 24 weeks and 48 weeks. HBeAg and anti-HBeAg will be examined at enrollment and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥20) with positive HBsAg who are prepared to receive systemic chemotherapy
* The presence of HBs antigen should be confirmed within recent two years
* The patients who could receive systemic chemotherapy in 4 weeks

Exclusion Criteria:

* Patients with poor performance status (Zubrod-ECOG ≥ 2 or Karnofsky score ≤ 70)
* Patients with cirrhosis
* Patients had eGFR lower than 15 ml/min/1.73m2 and didn't receive dialysis
* Patients had exposure to any NUC or interferon within 6 months before chemotherapy
* Patients were co-infected with HCV or HIV
* Allergy history to any tenofovir-based medication
* Pregnant woman
* Unable to sign inform consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of HBV reactivation during TAF prophylaxis | after 48 weeks of TAF use
  Definition of HBV reactivation :
  1. HBV DNA increase 2 log (100-fold) compared to the baseline level
  2. HBV DNA 3 log (1,000) IU/mL in a patient with previously undetectable level
  3. HBV DNA 4 log (10,000) IU/mL if the baseline level is not available

SECONDARY OUTCOMES:
The dynamic change of eGFR during TAF prophylaxis | after 48 weeks of TAF use
  record the dynamic change of eGFR from baseline to 48 weeks after TAF

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yueh Chen, MD, Principal Investigator — Ditmanson Medical Foundation Chiayi Christian Hospital
Locations (5):
- Taiwan (5):
  - Dalin Tzu Chi General Hospital, Chiayi City
  - Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City
  - St. Martin De Porress Hospital, Chiayi City
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Chi Mei Medical Hospital, Tainan

IPD SHARING:
Plan to Share IPD: No